CLINICAL TRIAL: NCT00412256
Title: Clinical Trial to Evaluate the Effect of Parenteral Supplementation With Omega-3-Fatty Acids in Patients With Rheumatoid Arthritis
Brief Title: Omegaven in Patients With Rheumatoid Arthritis (ORA-Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humanis Klinikum Niederosterreich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS4-EK-KAG/374
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2006-12-18 (Estimated); Status verified 2006-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Treatment; Disease activity; Clinical trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fish oil triglycerides

INTERVENTIONS:
Drug: Omegaven (10% fish-oil emulsion; Fresenius-Kabi)

SUMMARY:
The primary hypothesis constitutes that the fish-oil preparation (Omegaven) is superior to the preparation based on Soja-oil (Lipovenös)to reduce signs and symptoms in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
The study can be considered a phase III trial (comparison of two licensed preparations in a non-approved indication). This controlled double blind trial aims to compare the effect of parenterally applied fat emulsions on the disease activity of RA patients, as expressed by changes of the DAS28.

To test for the hypothesis patients are randomized and treated with 2ml/kg bodyweight of both preparations for seven consecutive days. These treatment cycles are repeated four times at monthly intervals. For not improving patients (DAS28 decrease <0.6) escapes before the third and the fourth treatment cycle are foreseen. In case of escape patients are treated with Omegaven in an open manner.

Efficacy parameters comprise the DAS28, the ACR-criteria, the M-HAQ, the SF-36, and the co-medication consumption. To assess safety laboratory parameters, comprising, LFT, KFT, CBC, fasting glucose, cholesterol, HDL, LDL, neutral fat, and urinary analysis are performed. Moreover, blood pressure control and clinically examinations are performed on a regular basis.

Study recruitment started in fall 2004 and was completed in November 2006.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* RA according to the ACR criteria
* active RA (DAS28 > 4.0) at the screening visit
* insignificant DAS28-change (<0.6) between screening and the first intervention

Exclusion Criteria:

* age lower than 18 yrs.
* pregnancy and insufficient birth control
* lactation
* army service
* lack of independence
* relevant therapeutic or dietary changes during the last three months
* relevant therapeutic or dietary changes foreseen for the study duration (including surgery)
* application of Omega-3 fatty acids during the last three months
* application of Omega-3 fatty acids intended for the study duration
* prednisolone > 10 mg/day
* contraindication for Omegaven or Lipovenös (according to the label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2006-11

PRIMARY OUTCOMES:
DAS28

SECONDARY OUTCOMES:
ACR-criteria, M-HAQ, VAS pain, SF-36,co-medication consumption

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard F Leeb, MD, Principal Investigator — Center for Rheumatology Lower Austria; Humanisklinikum NÖ
Locations (1):
- Center for Rheumatology Lower Austria, Humanisklinikum Lower Austria, Stockerau, Austria

REFERENCES:
- [Background] Leeb BF, Sautner J, Andel I, Rintelen B. Intravenous application of omega-3 fatty acids in patients with active rheumatoid arthritis. The ORA-1 trial. An open pilot study. Lipids. 2006 Jan;41(1):29-34. doi: 10.1007/11745-006-5066-x. PMID 16555468